### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for Exploration of the peripheral immune system in subjects with New Onset T1 Diabetes (NOT1D)

Compound Number : None

Effective Date : 09-Jun-2107

### **Description:**

• The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and outputs for the second interim analysis after the first 5 healthy volunteers (HVs) and 5 NOT1D subjects, The primary purpose of this interim analysis will be to facilitate decision making and study design for a potential follow-up interventional study.

#### **Author's Name and Functional Area:**

| PPD | | 07 Iva 2017 |
|----------------|-------------------------------|-------------|
| Principal Stat | istician, Clinical Statistics | 07-Jun-2017 |

### Approved by:

| PPD | | 09-Jun-2017 |
|-------------------|---------------------------------------|--------------|
| Director, Statist | cs & Programming, Clinical Statistics | 09-Juli-201/ |

Copyright 2016 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | <ul><li>2.1.</li><li>2.2.</li><li>2.3.</li></ul> | Change<br>Study O<br>Study D | KEY PROTOCOL INFORMATIONs to the Protocol Defined Statistical Analysis Planbjective(s) and Endpoint(s)sesign | 6<br>6<br>7 |
| | 2.4. | Statistic | al Hypotheses | 7 |
| 3. | PLANI<br>3.1. | | ALYSESAnalysesInterim Analysis 1 | 9 |
| | 3.2. | 3.1.2.<br>Final An | Interim Analysis 2alyses | |
| 4. | ANAL` | | PULATIONSI Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 11 |
| 6. | STUD<br>6.1. | | ATION ANALYSESw of Planned AnalysesInterim Analysis 1 | 12<br>12 |
| 7. | PRIMA<br>7.1. | | TISTICAL ANALYSES Ger Analyses Overview of Planned Biomarker Analyses 7.1.1.1. Interim Analyses 1 7.1.1.2. Interim Analyses 2 Planned Biomarker Statistical Analyses | 13<br>13<br>13 |
| 8. | SECO<br>8.1.<br>8.2. | Biomark<br>8.1.1. | STATISTICAL ANALYSES Arer Analyses Overview of Planned Biomarker Analyses Analyses Overview of Planned Adverse Event Analyses Overview of Planned Other Safety Analyses Interim Analysis 1 Interim Analysis 2 | 16<br>17<br>17<br>18 |
| 9. | REFE | RENCES | | 19 |
| 10. | APPE<br>10.2.<br>10.3. | Appendi<br>10.2.1.<br>Appendi<br>10.3.1. | ix 3: Data Display Standards & Handling Conventions | 22<br>22<br>24 |


# Clinical Study Identifier

| | | 10.3.2.1. | Baseline Definitions | 24 |
|---|---|---|---|---|
| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | 24 |
| | 10.3.3. | Reporting | Process & Standards | 24 |
| 10.4. | Appendix | k 4: Derive | d and Transformed Data | 26 |
| | 10.4.1. | | | |
| | 10.4.2. | Study Pop | oulation | 26 |
| | 10.4.3. | | | |
| 10.5. | Appendix | k 5: Premat | ture Withdrawals & Handling of Missing Data | 2 <mark>7</mark> |
| | 10.5.1. | Premature | e Withdrawals | <mark>27</mark> |
| | 10.5.2. | Handling of | of Missing Data | <mark>27</mark> |
| | | 10.5.2.1. | Handling of Missing Dates | <mark>27</mark> |
| | | 10.5.2.2. | | |
| | | 10.5.2.3. | Handling of Missing Data for Statistical | |
| | | | Analysis | 28 |
| 10.6. | Appendix | k 6: Values | of Potential Clinical Importance | |
| | 10.6.1. | Laborator | y Values | 29 |
| | 10.6.2. | | S | 30 |
| 10.7. | | | Checking and Diagnostics for Statistical | |
| | Analyses | 8 | | 31 |
| | 10.7.1. | Statistical | Analysis Assumptions | 31 |
| 10.8. | Appendix | | ker Analyses | |
| | 10.8.1. | | y of Leukocytes | 32 |
| | 10.8.2. | | y and phenotype of leukocyte subsets by flow | |
| | | cytometry | | 32 |
| | | | B_DC_Monocyte Panel | |
| | | | T Cell panel | |
| | | | Treg panel | |
| | | 10.8.2.4. | | |
| 10.9. | | | riations & Trade Marks | |
| | 10.9.1. | | ons | |
| | 10.9.2. | | ks | |
| 10.10. | | | f Data Displays | |
| | | | lay Numbering | |
| | | | mple Shell Referencing | |
| | | | e [Priority] | |
| | | | Tables | |
| | | | r Figures | |
| 10.11 | | | _istings | |
| 10.11. | Appendix | < 11: | ple Mock Shells for Data Displays | 41 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and outputs for the second interim analysis after the first 5 healthy volunteers (HVs) and 5 NOT1D subjects, the primary purpose of this interim analysis will be to facilitate decision making and study design for a potential follow-up interventional study. |
| Protocol | This RAP is based on the protocol amendment 3 (Dated: 07-Mar-2017) of study OTX203158 (GSK Document No.: 2015N246275_03] and eCRF Version 1.0. |
| Primary<br>Objective /<br>Endpoint | <ul> <li>To assess the frequency and phenotype of leukocyte subsets in iLN biopsies and peripheral blood in HVs and NOT1D subjects, measured by: <ul> <li>Absolute number and/or proportion of leukocyte subset in iLN biopsies and peripheral blood.</li> </ul> </li> </ul> |
| Secondary<br>Objectives /<br>Endpoint | To assess the frequency and phenotype of leukocyte subsets in iLN core biopsies and iLN fine needle aspirates in HVs and NOT1D subjects measured by: |
| | <ul> <li>To assess the safety and tolerability of iLN biopsy as well as expectations and experience of the biopsy procedure.</li> <li>Number of AEs and SAEs following lymph node biopsy procedure.</li> <li>Descriptive data obtained by a questionnaire on the acceptability of iLN biopsy in research setting.</li> </ul> |
| Study<br>Design | • A non-drug treatment study to compare differences in immune cells derived from iLN and peripheral blood of NOT1D subjects and HVs. Up to 15 evaluable NOT1D subjects and up to 15 evaluable HVs will be enrolled. The first interim analysis will assess the first 5 HVs, so as to determine the quality and quantity of cells. The second interim will assess the first 5 HVs and 5 NOT1D subjects Following the interim, for the remainder of the study the team will seek to match NOT1D subjects to HVs at a group level according to the number of subjects for each gender and the distribution of age within gender. |
| Planned<br>Analyses | Interim 1, Interim 2, Final |
| Analysis<br>Populations | Safety, Per Protocol, Core Biopsy, Fine Needle Aspirate Biopsy, Biopsy, Blood |
| Hypothesis | There are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives. |
| Primary<br>Analyses | The absolute values and proportion of flow cytometry cell counts of the iLN Biopsies and peripheral blood will be analyzed using generalized linear mixed models adjusting for group, sample type and the interaction of group and sample type. The model will include a subject random effect. |


# Clinical Study Identifier

| Overview | Key Elements of the RAP |
|---|---|
| Secondary<br>Analyses | <ul> <li>As per primary using only iLN Biopsy.</li> <li>In addition, safety data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.</li> </ul> |
| Exploratory<br>Analyses | <ul> <li>For this RAP, no exploratory endpoints will be described and details will be<br/>provided in subsequent RAPs.</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 3 (Dated: 06-Mar-2017).

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the frequency and phenotype of leukocyte subsets in iLN and peripheral blood in HVs and NOT1D subjects | Absolute number and/or proportion of leukocyte subsets in iLN and peripheral blood |
| Secondary Objectives | Secondary Endpoints |
| To assess the frequency and phenotype of leukocyte subsets in iLN core biopsies and iLN fine needle aspirates in HVs and NOT1D subjects | Absolute number and/or proportion of leukocyte subsets<br>in iLN core biopsies and iLN fine needle aspirates |
| To assess the safety and tolerability of iLN biopsy as well as expectations and experience of the biopsy procedure | <ul> <li>Number of AEs and SAEs following lymph node biopsy procedure</li> <li>Descriptive data obtained by a questionnaire on the</li> </ul> |
| | acceptability of iLN biopsy in research setting. |
| Exploratory Objectives* | Exploratory Endpoints |
| To assess suppression activity of T regulatory lymphocytes from the iLN and peripheral blood in HVs and NOT1D subjects | <ul> <li>Relative levels of T lymphocyte suppressive activity of<br/>cells from iLN and peripheral blood respectively</li> </ul> |
| To assess the frequency of cytokine-<br>producing lymphocytes in HVs and<br>NOT1D subjects | <ul> <li>Proportion of lymphocyte populations producing pro-<br/>inflammatory and/or anti-inflammatory cytokines in iLN<br/>and peripheral blood</li> </ul> |
| To assess clonal expansion of T and B lymphocyte populations in HVs and NOT1D subjects | Comparison of TCR and BCR usage in lymphocytes in iLN and peripheral blood |
| To assess the gene expression fingerprint of auto-antigen specific lymphocytes in HVs and NOT1D subjects | Gene expression levels of sorted auto antigen stimulated T lymphocyte populations in iLN and peripheral blood |
| 5) To assess the phenotype and transcriptomic fingerprint of stromal cells from iLN core biopsy samples in HVs and NOT1D subjects | Absolute number and/or proportion of stromal cell subsets and gene expression levels of stromal cell subsets from iLN core biopsy samples Stromal cell subsets Stromal cell s |

<sup>\*</sup> The Exploratory objectives / endpoints are listed in order of priority and the conduct of any experimental assays will be dependent on the material available (i.e. number of cells obtained) from iLN biopsies and peripheral blood.

### 2.3. Study Design



# 2.4. Statistical Hypotheses

This study is designed to explore the phenotype of immune cells in the iLN and peripheral blood (such as, but not restricted to PBMCs) of NOT1D subjects compared to HVs.

There are no formal hypotheses being tested due to the exploratory nature of the study. Primary comparisons of NOT1D subjects to HVs will be made using an estimation approach, providing point estimates and confidence intervals.

Secondary comparisons of biopsy methods will be made within NOT1D subjects and HVs using an estimation approach:

- iLN biopsies will be carried out by two related methods, fine-needle aspirate (FNA) and core biopsy sampling:
- If sufficient numbers of cells to meet the cell number requirements of the primary endpoint are obtained by both biopsy methods, the primary endpoint analysis will

be carried out independently for each biopsy method, otherwise only the biopsy method for which sufficient numbers of cells were obtained will be used for primary analysis.

- If no meaningful differences between biopsy methods are observed, material from both biopsy methods may be pooled to meet exploratory objectives 1, 2, 3 and 4. Material from fine-needle aspirate and core biopsies will not be pooled unless supported by the comparison described above.
- If meaningful differences in the proportion of leukocyte subsets between cells derived from each biopsy method are observed, then:
  - o If sufficient number of core biopsy derived cells are available, these will be analysed for exploratory objectives 1 and 2.
  - o Fine needle aspirate derived cells will be used to meet exploratory objectives 3 and 4. If insufficient number of core biopsy derived cells are available to meet exploratory objectives 1 and 2, then fine needle aspirate derived cells may be used to meet either or both of those exploratory objectives.

A graphical representation of the comparisons are shown in Figure 1.



Figure 1 - Graphical representation of comparisons

### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

### 3.1.1. Interim Analysis 1

A data look will be carried after the recruitment of a cohort of up to 5 HVs to determine if the quality and quantity of cells derived from either fine needle aspirate or core biopsy of the inguinal lymph node and from peripheral blood are likely to be sufficient to continue the study to meet its primary objective.

The decision rules for the study to continue are:

- Peripheral blood yields  $> 1 \times 10e^6$  cells, and
- Yield from either iLN biopsy samples  $> 1 \times 10e^6$  cells.

In addition, the data from the interim analysis will be used to explore the assumptions and feasibility of the primary statistical analysis, and may also be used for pre-programming of outputs for the final analysis.

If the decision is taken to stop the study at the interim, the full safety outputs plus listings of other collected data will be produced.

# 3.1.2. Interim Analysis 2

An interim analysis will be carried out after the recruitment of 5 evaluable HVs and 5 evaluable NOT1D subjects. The primary purpose of this interim analysis will be to facilitate decision making and study design for a potential follow-up interventional study.

In addition, the interim analysis results would also help to enable prioritization of the exploratory assays and to facilitate the final RAP. Due to uncertainty around variability and precision, the primary analyses described in Section 7 will be performed in order to re-assess the precision of estimates for the comparisons of interest.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | Comprised of all subjects who complete any | <ul> <li>Study Population</li> </ul> |
| | study assessment | <ul> <li>Safety</li> </ul> |
| Core Biopsy | Subjects in the 'Safety' population for whom at least one lymph node core biopsy was taken | Biomarker |
| Fine needle aspirate Biopsy | Subjects in the 'Safety' population for whom at least one lymph node fine needle aspirate biopsy was taken | Biomarker |
| Biopsy | Subjects in both 'Core Biopsy' and 'fine needle aspirate biopsy' populations | Biomarker |
| Blood | Subjects in the 'Safety' population for whom one blood sample was taken for analysis of cells derived from peripheral blood. | Biomarker |
| Per Protocol | Subjects in the 'Safety' Population who were compliant with the Protocol | Biomarker |

#### NOTES:

- Please refer to
- Appendix 10: List of Data Displays which details the population to be used for each displays being generated.

### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP).
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.
- Analyses may be repeated on the Per Protocol population if deemed important.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

There are planned examination of covariates and subgroups.

There are no planned adjustments made for multiple centres in this study.

There are no planned adjustments for multiple comparisons or multiplicity.

### Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | |
| | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Model Checking and Diagnostics for Statistical Analyses |
| 10.8 | Appendix 8: Biomarker Analyses |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays

Table 2 Overview of Planned Study Population Analyses

| Endpoint / Parameter / Display Type | Data I | Data Displays Generated | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition | Y | | |
| Reasons for Screen Failure | Υ | | Υ |
| Subjects by Country and Centre | Y | | |
| Reasons for Subject Withdrawal | | | Υ |
| Protocol Deviations | | | |
| Important Protocol Deviations | | | Υ |
| Subjects with Inclusion/Exclusion Criteria Deviations | | | Υ |
| Populations Analysed | | | |
| Study Populations and Exclusions | Y | | |
| Subjects Excluded from Any Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Race and Racial Combinations | Y | | Υ [1] |
| Race and Racial Combination Details | Y | | |
| Prior and Concomitant Medications | | | |
| Past Medical Conditions | Y | | |
| Concomitant Medications | Y | | Υ |

### NOTES:

[1] Listing of race.

### 6.1.1. Interim Analysis 1

No study population analyses will be produced for the first interim analysis.

### 6.1.2. Interim Analysis 2

No study population analyses will be produced for the first interim analysis.

<sup>•</sup> Y = Yes display generated.


Clinical Study Identifier

### 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Biomarker Analyses

### 7.1.1. Overview of Planned Biomarker Analyses

The primary biomarker analyses will be based on the 'Safety' population, unless otherwise specified.

Between group (HV vs NOT1D) comparisons will use data from all subjects who have at least one evaluable sample from either method. Between method comparisons and analyses will only be performed in subjects who provide sufficient cells from both methods in each pairwise comparison (as shown in Figure 1).

If sufficient numbers of cells to meet the cell number requirements of the primary endpoint are obtained by both biopsy methods, the primary endpoint analysis will be carried out independently for each biopsy method, otherwise only the biopsy method for which sufficient numbers of cells were obtained will be used for primary analysis.

Table 3 provides an overview of the planned biomarker analyses, with full details of data displays being presented in

Appendix 10: List of Data Displays.

Table 3 Overview of Biomarker Analyses

| Endpoint | Absolute | | | | | | | | Proportion | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Stats Analysis | | | Summary Ir | | Individual Stats Ana | | s Anal | ysis | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | Г |
| iLN Biopsies and Peripheral Blood | | | | | | | | | | | | | | |
| Leukocyte subsets | eukocyte subsets Y Y | | | | | | Υ | Υ | | Υ | Υ | Y | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 7.1.1.1. Interim Analyses 1

The analysis performed at the interim will be a subset of the final analysis as given by Table 4.

Table 4 Overview of Biomarker Analyses for Interim

| Endpoint | | Absolute | | | | | | Proportion | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis S | | Sum | Summary Individual | | Stats Analysis | | ysis | Summary | | Individual | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| iLN Biopsy and Peripheral Blood | | | | | | | | | | | | | | |
| Leukocyte Count | | | | Υ | | | Υ | | | | | | | |

#### NOTES:

• T = Table, F = Figure, L = Listing, Y = Yes display generated.

| Endpoint | Absolute | | | | | Proportion | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis Sumn | | mary | Indiv | idual | Stats Analysis | | Summary | | Individual | | | | |
| | Т | F | L | Τ | F | F | L | Τ | F | L | Τ | F | F | L |

- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 7.1.1.2. Interim Analyses 2

The analysis performed at the interim will be a subset of the final analysis as given by Table 4.

### Table 5 Overview of Biomarker Analyses for Interim

| Endpoint | | Absolute | | | | | | Proportion | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis S | | Summary Individual | | Stats Analysis | | ysis | Summary | | Individual | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | Г |
| iLN Biopsy and Peripheral Blood | | | | | | | | | | | | | | |
| Leukocyte Count | | | | Υ | | | Υ | Υ | Υ | | Υ | Υ | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 7.1.2. Planned Biomarker Statistical Analyses

### **Primary Statistical Analyses**

### Endpoint(s)

Proportion of flow cytometry cell counts

### **Model Specification**

- Endpoints analyzed for each flow cytometry cell type using generalized linear mixed models (GLMM).
- The analysis will be performed on the parameters listed in Appendix 8: Biomarker Analyses
- Terms in GLMM model will include:

Fixed categorical: group, sample type, and the interaction of group with sample type Random effect: subject

Where group is either HV or NOT1D, and sample type is peripheral blood, core biopsy or fine needle aspirate.

### **Model Checking & Diagnostics**

• Refer to Appendix 7: Model Checking and Diagnostics for Statistical Analyses

### **Model Results Presentation**

 For proportional cell counts, these models will estimate the mean (or geometric) cell count for each sample type in each group, comparing means using ratios as outlined in the primary hypothesis section.

# 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Biomarker Analyses

# 8.1.1. Overview of Planned Biomarker Analyses

As per Primary Analysis, see Section 7.1.2, but for secondary comparisons detailed in Figure 1.

# 8.2. Safety Analyses

### 8.2.1. Overview of Planned Adverse Event Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in

Appendix 10: List of Data Displays.

Table 6 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Absol | ute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | T | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC | Υ | | Υ |
| Common AEs by Overall Frequency | Υ | | |
| Common Grade 2-4 AEs by Overall Frequency | Υ | | |
| Subjects & No. of Occurrences of Common Non-Serious AEs by SOC and PT | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs | Υ | | Υ |
| Non-Fatal Serious AEs | | | Υ |
| Serious AEs by SOC | Υ | | |
| Reasons for Considering as a Serious AE | | | Υ |
| AEs Leading to Withdrawal from Study by Overall Frequency | Υ | | Y |
| Subjects and Number of Occurrences of Serious and Fatal Serious AEs | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.2.2. Overview of Planned Other Safety Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in

Appendix 10: List of Data Displays.

Table 7 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Summary Individual | | Summary | | Individual | |
| | Т | F | L | Т | F | L |
| Laboratory Values | | | | | | |
| Haematology | | | Y | | | |
| Clinical Chemistry | | | Y | | | |
| Urinalysis | | | Y | | | |
| Other Screening Tests | | | Y | | | |
| Vital Signs | | | | | | |
| Vitals Findings | Υ | | Y | Υ | | Υ |
| Vitals Values (PCI) | Υ | | Y | | | |

### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.2.3. Interim Analysis 1

No formal safety analyses will be produced for the interim analysis.

### 8.2.4. Interim Analysis 2

No formal safety analyses will be produced for the interim analysis.

# 9. REFERENCES

GlaxoSmithKline Document Number 2015N246275\_03 (2017-MAR-06 Amendment No. 3): Exploration of the peripheral immune system in subjects with New Onset T1 Diabetes (NOT1D)

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| Section 10.2 | |
| | Appendix 2: Time & Events |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Biomarkers |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Model Checking and Diagnostics for Statistical Analyses |
| Section 10.8 | Appendix 8: Biomarker Analyses |
| Other RAP | |
| Appendices | |
| Section 10.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 10.10 | Appendix 10: List of Data Displays |
| Section 10.11 | Appendix 11: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 10.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|--------|----------------------------------------|
| 01 | Eligibility criteria not met |
| 02 | Excluded medication, vaccine or device |
| 03 | Equipment procedures |
| 04 | Biological sample specimen procedures |

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Events

Screening procedures in addition to those listed below are (outpatient visit): Informed consent; Inclusion / Exclusion criteria; demography.

| Procedure | Screening (between -<br>42 to 7 days prior to<br>study session) | | | Telephone<br>follow-up<br>Day ~2 to<br>~ Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes | |
|---|---|---|---|---|---|---|---|
| | | Pre biopsy | Biopsy | End of study<br>session visit | | | |
| Full physical<br>exam | х | | | | | | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Medical history /<br>Past and current<br>medical<br>conditions | х | | | | | | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Laboratory<br>assessments (see<br>Section 6.7.5) | x | | | | | | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Concomitant<br>medication<br>review | х | X | | | X | x | , |
| Alcohol Urine<br>Test and Test for<br>Drugs of Abuse | X | X | | | | | |

| Procedure | Screening (between -<br>42 to 7 days prior to<br>study session) | | Study Session Day 1 | | Notes |
|---|---|---|---|---|---|
| | | Pre biopsy | Biopsy | End of study<br>session visit | |
| Urine Pregnancy<br>test (in women of<br>child bearing<br>potential) | х | х | | | |
| Vital signs | х | х | | х | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Medical history /<br>Past and current<br>medical<br>conditions | | X | | | |
| Proposed biopsy<br>site review | | X | | | |
| Peripheral blood<br>collection for<br>cell isolation and<br>metabonomics<br>analyses | | х | | | |
| Peripheral blood<br>collection for<br>genetics | | X | | | |


# Clinical Study Identifier

| Procedure | Screening (between -<br>42 to 7 days prior to<br>study session) | | | Telephone<br>follow-up<br>Day ~2 to<br>~ Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes | |
|---|---|---|---|---|---|---|---|
| | | Pre biopsy | Biopsy | End of study<br>session visit | | | |
| Peripheral blood<br>collection for<br>haematology,<br>clinical<br>chemistry only,<br>(see Section<br>6.7.5) | | х | | | | | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Inguinal lymph node biopsy (fine needle aspirate & core biopsy) | | | х | | | | |
| Wound<br>assessment | | | | x | X<br>(telephone) | X<br>(telephone | To be completed if a<br>post study visit is<br>required. Attendance to<br>the unit post study<br>sessions only if<br>necessary (at discretion<br>of investigator) |
| Pre- & post-<br>biopsy<br>questionnaire to<br>assess subject<br>experience of<br>lymph node<br>biopsy | | х | | | X<br>(via<br>telephone:<br>questionnai<br>re to be<br>filled in on<br>the day<br>after the<br>procedure) | | |

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

# 10.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| Α | No Treatment | No Treatment | 1 |

### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

| | Study Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| 1 | Healthy Volunteers | Healthy Volunteers | 1 |
| 2 | NOT1D | NOT1D | 2 |

### 10.3.2. Baseline Definition & Derivations

### 10.3.2.1. Baseline Definitions

For all endpoints the baseline value will be the latest pre-biopsy assessment.

### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | =Post-Biopsy Value – Baseline |
| % Change from Baseline | =100 x [(Post-Biopsy Value – Baseline) / Baseline] |

### 10.3.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently sugerneration of discrete. | pported versions of SAS software will be used to perform all data analyses and splays. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : \\arprod\nocompound\mid203158\[reporting effort] |
| | \\arwork\nocompound\mid203158\[reporting effort] |
| QC Spreadsheet | : \\arprod\nocompound\mid203158\[reporting effort]\qc |
| <b>Analysis Datasets</b> | |

### **Reporting Process**

• Analysis datasets will be created according to Legacy GSK A&R dataset standards.

### **Generation of RTF Files**

RTF files will be generated for the final analysis only.

### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - RTF files will be generated for displays

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

#### **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|------------------|--------------------------------------------|
| Categorical Data | N, n, frequency, % |

## 10.4. Appendix 4: Derived and Transformed Data

### 10.4.1. **General**

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from date of biopsy :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Biopsy Date → Study Day = Ref Date Biopsy Date</li>
  - Ref Data ≥ Biopsy Date → Study Day = Ref Date (Biopsy Date) + 1

### 10.4.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

### 10.4.3. Safety

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined one who has completed all phases of the study including the follow-up call(s). The end of the study is defined as the last subject's last telephone call As defined in the protocol the overall study duration for each subject will be up to 8 weeks, including the screening period.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in displays, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

Completely missing dates will remain missing, with no imputation applied

### 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day</li> </ul> |
| | (dependent on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |

# 10.5.2.3. Handling of Missing Data for Statistical Analysis

Missing data will remain missing with no imputation applied for the purposes of statistical analysis.

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) High Flag (>x | |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | <b>↑ 44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte Units Category Clinical Concern Rang | | | |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower Upper | |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

# 10.7. Appendix 7: Model Checking and Diagnostics for Statistical Analyses

### 10.7.1. Statistical Analysis Assumptions

| Endpoint(s) | • | Proportion of flow cytometry cell counts |
|-------------|---|------------------------------------------|
| Analysis | • | GLMM |

- Model assumptions will be applied, but appropriate adjustments maybe applied based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the RANDOM line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

# 10.8. Appendix 8: Biomarker Analyses

# 10.8.1. Frequency of Leukocytes

| Test Analyte | Details |
|---|---|
| Core biopsy total cell number | Total number of cells obtained from pooled core biopsies |
| Fine Needle Aspirate total cell number | Total number of cells obtained from pooled fine needle aspirates |

# 10.8.2. Frequency and phenotype of leukocyte subsets by flow cytometry

# 10.8.2.1. B\_DC\_Monocyte Panel

| Test Analyte | Details |
|---|---|
| %DC (MNC) | NONCD16hiCD3-CD19-HLADR+CD14-CD16- |
| %Myeloid DC (DC) | NONCD16hiCD3-CD19-CD14-CD16-HLADR+CD11C+CD123- |
| %pDC (DC) | NONCD16hiCD3-CD19-CD14-CD16-HLADR+CD11C-CD123+ |
| %Plasmablast (B) | NONCD16hiCD19+CD27+CD38+ |
| %Circulating B (B) | NONCD16hiCD19+Plasmablast-CD27+lgD+ |
| %Classical B (B) | NONCD16hiCD19+Plasmablast-CD27+lgD- |
| %Double neg B (B) | NONCD16hiCD19+Plasmablast-CD27-lgD- |
| %Naïve B (B) | NONCD16hiCD19+Plasmablast-CD27-lgD+ |
| %Transitional B (B) | NONCD16hiCD19+Plasmablas-CD27-lgD+CD38+CD24+ |
| %CD56bright NK (NK) | NONCD16hiCD3-CD19-CD14-CD16-CD56hi |
| %CD56loCD16+ NK (NK) | NONCD16hiCD3-CD19-CD14-CD56loCD16+ |
| %CD56loCD16- NK (NK) | NONCD16hiCD3-CD19-CD14-CD56loCD16- |
| %CD14+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD14+ |
| %CD14+CD16+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD14+CD16+ |
| %CD16+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD16+ |

# 10.8.2.2. T Cell panel

| Test Analyte | Details |
|----------------------|----------------------------|
| %CD8 Tn (CD8) | CD3+CD4-CD45RA+CCR7+CD95- |
| %CD8 Tcm (CD8) | CD3+CD4-CD45RA-CCR7+ |
| %CD8 Tem (CD8) | CD3+CD4-CD45RA-CCR7- |
| %CD8 Temra (CD8) | CD3+CD4-CD45RA+CCR7- |
| %CD8 Tscm (CD8) | CD3+CD4-CD45RA+CCR7+CD95+ |
| %Tconv Tn (Tconv) | CD4+Treg-CD45RA+CCR7+CD95- |
| %Tconv Tcm (Tconv) | CD4+Treg-CD45RA-CCR7+ |
| %Tconv Tem (Tconv) | CD4+Treg-CD45RA-CCR7- |
| %Tconv Temra (Tconv) | CD4+Treg-CD45RA+CCR7- |

| Test Analyte | Details |
|---|---|
| %Tconv Tscm (Tconv) | CD4+Treg-CD45RA+CCR7+CD95+ |
| %Tconv Th1 (mTconv) | CD4+Treg-CXCR5-CXCR3+CCR10-CCR6- |
| %Tconv Th1Th17 (mTconv) | CD4+Treg-CXCR5-CXCR3+CCR10-CCR6+ |
| %Tconv Th17 (mTconv) | CD4+Treg-CXCR5-CXCR3-CCR4+CCR10-CCR6+ |
| %Tconv Th2 (mTconv) | CD4+Treg-CXCR5-CXCR3-CCR4+CCR10-CCR6- |
| %Tconv Th22 (mTconv) | CD4+Treg-CXCR5-CXCR3-CCR4+CCR10+CCR6+ |
| %Tconv Tfh (mTconv) | CD4+Treg-CXCR5+ |
| %Tconv PD-1+ ICOS+ Tfh (mTconv) | CD4+Treg-CXCR5+PD-1+ICOS+ |
| %Treg Th1 (mTreg) | CD4+CD25+CD127loCXCR5-CXCR3+CCR10-CCR6- |
| %Treg Th1Th17 (mTreg) | CD4+CD25+CD127loCXCR5-CXCR3+CCR10-CCR6+ |
| %Treg Th17 (mTreg) | CD4+CD25+CD127loCXCR5-CXCR3-CCR4+CCR10-CCR6+ |
| %Treg Th2 (mTreg) | CD4+CD25+CD127loCXCR5-CXCR3-CCR4+CCR10-CCR6- |
| %Treg Th22 (mTreg) | CD4+CD25+CD127loCXCR5-CXCR3-CCR4+CCR10+CCR6+ |
| %Treg Tfh (mTreg) | CD4+CD25+CD127loCXCR5+ |
| %Treg PD-1+ ICOS+ Tfh (mTreg) | CD4+CD25+CD127loCXCR5+PD-1+lCOS+ |

# 10.8.2.3. Treg panel

| Test Analyte | Details |
|--------------------------|-----------------------------------|
| %CD15s+ Tconv (Tconv) | CD3+CD4+CD25-FOXP3-CD15S+ |
| %CD69+ Tconv (Tconv) | CD3+CD4+CD25-FOXP3-CD69+ |
| %Helios+ Tconv (Tconv) | CD3+CD4+CD25-FOXP3-HELIOS+ |
| %Ki67+ Tconv (Tconv) | CD3+CD4+CD25-FOXP3-KI67+ |
| %CD15s+ mTconv (mTconv) | CD3+CD4+CD25-FOXP3-CD45RA-CD15S+ |
| %CD69+ mTconv (mTconv) | CD3+CD4+CD25-FOXP3-CD45RA-CD69+ |
| %Helios+ mTconv (mTconv) | CD3+CD4+CD25-FOXP3-CD45RA-HELIOS+ |
| %Ki67+ mTconv (mTconv) | CD3+CD4+CD25-FOXP3-CD45RA-KI67+ |
| %Treg (CD4) | CD3+CD4+CD25+FOXP3+ |
| %aTreg (Treg) | CD3+CD4+CD25+FOXP3+CD45RA- |
| %mTreg (Treg) | CD3+CD4+CD25+FOXP3medCD54RA- |
| %rTreg (Treg) | CD3+CD4+CD25+FOXP3medCD45RA+ |
| %CD15s+ Treg (Treg) | CD3+CD4+CD25+FOXP3+CD15S+ |
| %CD69+ Treg (Treg) | CD3+CD4+CD25+FOXP3+CD69+ |
| %Helios+ Treg (Treg) | CD3+CD4+CD25+FOXP3+HELIOS+ |
| %Ki67+ Treg (Treg) | CD3+CD4+CD25+FOXP3+KI67+ |
| %CD69+ CD8 (CD8) | CD3+CD8+CD69+ |
| %Ki67+ CD8 (CD8) | CD3+CD8+KI67+ |

# CONFIDENTIAL

# 10.8.2.4. Suppressive activity of regulatory cells

| Test Analyte | Details |
|----------------------------|------------------------------------|
| Percentage suppression 0:1 | Treg: Tconventional cell ratio 0:1 |
| Percentage suppression 1:2 | Treg: Tconventional cell ratio 1:2 |
| Percentage suppression 1:4 | Treg: Tconventional cell ratio 1:4 |

# 10.9. Appendix 9: Abbreviations & Trade Marks

# 10.9.1. Abbreviations

| Abbreviation | Description |
|--------------|-------------------------------------------|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| BL | Baseline |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FNA | Fine needle aspirate |
| HV | Healthy volunteer |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| iLN | Inguinal lymph node |
| IMMS | International Modules Management System |
| GLMM | Generalized linear mixed model |
| GUI | Guidance |
| GSK | GlaxoSmithKline |
| NOT1D | New Onset Type 1 Diabetes Mellitus |
| PBMC | Peripheral blood mononuclear cell |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| PT | Preferred Term |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SOC | System Organ Class |
| TCR / BCR | T-cell Receptor / B-cell Receptor |
| TFL | Tables, Figures & Listings |
## 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| | SAS |

## 10.10. Appendix 10: List of Data Displays

#### 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|--------------|--------------|
| Study Population | 1.01 to 1.nn | 1.01 to 1.nn |
| Safety | 2.01 to 2.nn | 2.01 to 2.nn |
| Pharmacodynamic and / or Biomarker | 3.01 to 3.nn | 3.01 to 3.nn |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.10.3. Deliverable [Priority]

| Delivery | Description |
|----------|------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |

## 10.10.4. Biomarker Tables

| Bion | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| Freq | uency and | d phenotype | e of leukocyte subsets by flow cytometry | | |
| 3.1. | Safety | PD_T1 | Summary of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3.2. | Safety | PD_T2 | Statistical Analyses of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3.3. | Safety | PD_T1 | Summary of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC |
| 3.4. | Safety | PD_T2 | Statistical Analyses of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC |
| 3.5. | Safety | PD_T1 | Summary of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC |
| 3.6. | Safety | PD_T2 | Statistical Analyses of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC |
| Supp | Suppressive activity of regulatory cells | | | | |
| 3.7. | Safety | PD_T1 | Summary of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC |
| 3.8. | Safety | PD_T2 | Statistical Analyses of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC |

## 10.10.5. Biomarker Figures

| Bion | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| Freq | Frequency and phenotype of leukocyte subsets by flow cytometry | | | | |
| 3.1. | Safety | PD_F1 | Boxplots of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3.2. | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of B_DC_Monocyte Panel | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3.3. | Safety | PD_F1 | Boxplots of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC |
| 3.4. | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of T Cell Panel | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3.5. | Safety | PD_F1 | Boxplots of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC |
| 3.6. | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of Treg Panel | Parameters listed in Section 10.8.2.1 | IA SAC |
| Supp | Suppressive activity of regulatory cells | | | | |
| 3.7. | Safety | PD_F1 | Boxplots of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC |
| 3.8. | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of Suppressive activity of regulatory cells | Parameters listed in Section 10.8.2.1 | IA SAC |

## 10.10.6. Non-ICH Listings

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| Freq | uency and | d phenotype | e of leukocyte subsets by flow cytometry | | |
| 1. | Safety | PD_L1 | Listing of B_DC_Monocyte Panel by Biomarker | Parameters listed in Section 10.8.2.1 | IA SAC |
| 2. | Safety | PD_L2 | Listing of B_DC_Monocyte Panel by Group and Subject ID | Parameters listed in Section 10.8.2.1 | IA SAC |
| 3. | Safety | PD_L1 | Listing of T Cell Panel by Biomarker | Parameters listed in Section 10.8.2.2 | IA SAC |
| 4. | Safety | PD_L2 | Listing of T Cell Panel by Group and Subject ID | Parameters listed in Section 10.8.2.2 | IA SAC |
| 5. | Safety | PD_L1 | Listing of Treg Panel by Biomarker | Parameters listed in Section 10.8.2.3 | IA SAC |
| 6. | Safety | PD_L2 | Listing of Treg Panel by Group and Subject ID | Parameters listed in Section 10.8.2.3 | IA SAC |
| Sup | Suppressive activity of regulatory cells | | | | |
| 7. | Safety | PD_L1 | Listing of Suppressive activity of regulatory cells by Biomarker | Parameters listed in Section 10.8.2.4 | IA SAC |
| 8. | Safety | PD_L2 | Listing of Suppressive activity of regulatory cells by Group and Subject ID | Parameters listed in Section 10.8.2.4 | IA SAC |

## 10.11. Appendix 11: Example Mock Shells for Data Displays

## Example: PD\_T1


Population: Safety

Method

Subset: XXXXXXXXX (Unit)

| | | | | Method | |
|-------|----|-----------|--------------|--------------|--------------|
| Group | N | Statistic | Blood | FNA | Core |
| HV | XX | n | XX | XX | XX |
| | | Mean (SD) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | | 95% CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | | Min | X.X | X.X | X.X |
| | | Median | X.XX | X.XX | X.XX |
| | | Max | X.X | X.X | X.X |
| NOT1D | XX | n | XX | XX | XX |
| | | Mean (SD) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | | 95% CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | | Min | X.X | X.X | X.X |
| | | Median | X.XX | X.XX | X.XX |
| | | Max | X.X | X.X | X.X |

Note: n is the number of subjects with evaluable data for the specific biopsy.

203158

#### Example: PD\_T2 - Page 1


Population: Safety

Table X.X Statistical Analyses of XXXXX by Method and Patient Group

Group

Subset: XXXXXXXXX (Unit)

| | | | Group | |
|---|---|---|---|---|
| Method | Statistic | HV (N=XX) | NOT1D (N=XX) | Difference |
| Blood | n | XX | XX | |
| | LS Mean (SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | 95% CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| iLN | n | XX | XX | |
| | LS Mean (SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | 95% CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| FNA | n | XX | XX | |
| | LS Mean (SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | 95% CI | x.xx, x.xx | X.XX, X.XX | X.XX, X.XX |
| Core | n | XX | XX | |
| 0010 | LS Mean (SE) | X.XX (X.XXX) | X.XX (X.XXX) | X.XX (X.XXX) |
| | 95% CI | X.XX, X.XX | X.XX, X.XX | X.XX, X.XX |
| | JJ 0 CI | $\Lambda \cdot \Lambda \Lambda_{I} \Lambda \cdot \Lambda \Lambda$ | $\Lambda \cdot \Lambda \Lambda / \Lambda \cdot \Lambda \Lambda$ | $\Lambda \cdot \Lambda \Lambda_{I} \Lambda \cdot \Lambda \Lambda$ |

Note: n is the number of subjects with evaluable data for the specific biopsy. Only subjects with data for both pairs of methods will be used in the comparisons. Model used...

#### Example: PD\_T2 - Page 2


Population: Safety

Table X.X Statistical Analyses of XXXXX by Method and Patient Group

Subset: XXXXXXXXX (Unit)

| | • | | Group |
|---|---|---|---|
| Comparison | Statistic | HV (N=XX) | NOT1D (N=XX) |
| iLN vs Blood | n | XX | XX |
| | LS Mean (SE) - iLN | X.XX (X.XXX) | X.XX (X.XXX) |
| | LS Mean (SE) - Blood | X.XX (X.XXX) | X.XX (X.XXX) |
| | LS Mean Ratio (95% CI) | X.XX (X.XX, X.XX) | X.XX (X.XX, X.XX) |
| FNA vs Blood | n | XX | XX |
| | LS Mean (SE) - iLN | X.XX (X.XXX) | X.XX (X.XXX) |
| | LS Mean (SE) - Blood | X.XX (X.XXX) | X.XX (X.XXX) |
| | LS Mean Ratio (95% CI) | X.XX (X.XX, X.XX) | X.XX (X.XX, X.XX) |

. . . .

Continue for Core vs Blood

FNA vs Core

Note: n is the number of subjects with evaluable data for the specific biopsy. Only subjects with data for both pairs of methods will be used in the comparisons. Model used...

## Example: PD\_F1

Protocol: OTX203158 Population: Safety

Figure X.X
Boxplots of XXXXX by Method and Patient Group

Biomarker: XXXXXXXXX (Unit)




Protocol: OTX203158 Population: Safety

Figure X.X LS Mean Estimates and Differences with 95% CI of XXXXX

Biomarker: XXXXXXXXX (Unit)




Protocol: OTX203158 Population: Safety

Figure X.X LS Mean Estimates and Differences with 95% CI of XXXXX

Biomarker: XXXXXXXXX (Unit)




Protocol: OTX203158 Population: Safety

Figure X.X LS Mean Estimates and Differences with 95% CI of XXXXX

Biomarker: XXXXXXXXX (Unit)




203158

## Example: PD\_L1

Protocol: OTX203158

Page 1 of X

Population: Safety

Listing X

Listing of XXXXX by Biomarker

Biomarker: XXXXXXXXX (Unit)

| | | | | Metho | od |
|---|---|---|---|---|---|
| Group | Subje | ect ID/Age/Sex/Race | Blood | FNA | Core |
| HV | PPD | /XX/X/XXXXXXX<br>/XX/X/XXXXXXX<br>/XX/X/XXXXXX | X.X | | |
| NOT1D | | /xx/x/xxxxxxx<br>/xx/x/xxxxxxx<br>/xx/x/xxxxxx | | | |


203158

## Example: PD\_L2


Population: Safety

Group/Subject ID/Age/Sex/Race: HV PPD /XX/X/XXXXXXX

| | | Method | |
|-------------|-------|--------|------|
| Biomarker | Blood | FNA | Core |
| Biomarker 1 | X.X | X.X | X.X |
| Biomarker 2 | X.X | X.X | X.X |
| Biomarker 3 | X.X | X.X | X.X |
| Biomarker 4 | X.X | X.X | X.X |

•••

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title: Reporting and Analysis Plan for Exploration of the peripheral<br/>immune system in subjects with New Onset T1 Diabetes<br/>(NOT1D)Compound Number: NoneEffective Date: 15-JAN-2018

#### **Description:**

• The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and outputs for the final analyses.

#### **RAP Author(s):**

PPD

Statistics Leader (II Clinical Statistics)

#### The GlaxoSmithKline group of companies

#### **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Programmer (II Clinical Programming) | 12-JAN-2018 | PharmaTMF |
| Scientific leader (II DPU Mechanistic Medicine Discovery) | 15-JAN-2018 | Email |
| Manager Translational Medicine (II DPU Mechanistic Medicine Discovery) | 10-JAN-2018 | PharmaTMF |
| Data Quality Leader (II Clinical Pharmacology<br>Science and Study Operations) | 12-JAN-2018 | PharmaTMF |
| Principal Clinical Research Scientist (II Clinical Pharmacology Science and Study Operations) | 12-JAN-2018 | PharmaTMF |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|----------------------------------------------|-------------|-----------------|
| Statistics Director (II Clinical Statistics) | 12-JAN-2018 | PharmaTMF |
| Job Title (II Clinical Programming) | 12-JAN-2018 | PharmaTMF |

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 6 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 7 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| 3. | PLAN | NED ANALYSES | 10 |
| | 3.1. | Interim Analyses | |
| | | 3.1.1. Interim Analysis 1 | |
| | | 3.1.2. Interim Analysis 2 | |
| | 3.2. | Final Analyses | 10 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 11 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | /ENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Change from Baseline Definitions | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 13 |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5.<br>5.6. | Multiple Comparisons and Multiplicity | |
| | 5.0.<br>5.7. | Multiple Comparisons and Multiplicity Other Considerations for Data Analyses and Data Handling | 13 |
| | <b>U</b> | Conventions | 13 |
| _ | OTUD | NV DODIN ATION ANALYOFO | 4.4 |
| 6. | | OVER THE REPORT OF PROPERTY OF THE PROPERTY OF | |
| | 6.1. | Overview of Planned Analyses | |
| | | 6.1.1. Interim Analysis 1 | |
| | | 6.1.2. Interim Analysis 2 | 14 |
| 7. | PRIM | ARY STATISTICAL ANALYSES | 15 |
| | 7.1. | Biomarker Analyses | 15 |
| | | 7.1.1. Overview of Planned Biomarker Analyses | |
| | | 7.1.1.1. Interim Analyses 1 | |
| | | 7.1.1.2. Interim Analyses 2 | |
| | | 7.1.2. Planned Biomarker Statistical Analyses | |
| | 7.2. | Secondary statistical analyses | |
| | 7.3. | Biomarker Analyses | |
| | | 7.3.1. Overview of Planned Biomarker Analyses | 16 |
| 8. | | TY ANALYSES | |
| | 8.1. | Adverse Events Analyses | |
| | 8.2. | Clinical Laboratory Analyses | |
| | 8.3. | Other Safety Analyses | 17 |


| | | 8.3.1. | Interim Analysis 1 | |
|---|---|---|---|---|
| | | 8.3.2. | Interim Analysis 2 | 17 |
| 9. | REFE | RENCES. | | 18 |
| 40 | 4 DDE1 | UDIOFO | | 40 |
| 10. | | | A. Dark and Darking Management and Daffarition of a Dark | 19 |
| | 10.1. | | (1: Protocol Deviation Management and Definitions for Per | 40 |
| | | 10 1 1 | Population | 19 |
| | 10.2. | | Exclusions from Per Protocol Population | |
| | 10.2. | | Protocol Defined Time & Events | |
| | 10.3. | | 3: Data Display Standards & Handling Conventions | |
| | 10.5. | | Reporting Process | |
| | | 10.3.1. | | |
| | 10.4. | | (4: Derived and Transformed Data | |
| | | 10.4.1. | General | |
| | | 10.4.2. | Study Population | |
| | | 10.4.3. | Safety | |
| | 10.5. | Appendix | c 5: Premature Withdrawals & Handling of Missing Data | |
| | | 10.5.1. | | |
| | | 10.5.2. | Handling of Missing Data | |
| | | | 10.5.2.1. Handling of Missing Dates | 27 |
| | | | 10.5.2.2. Handling of Partial Dates | 27 |
| | | | 10.5.2.3. Handling of Missing Data for Statistical | |
| | | | Analysis | 28 |
| | 10.6. | | c 6: Values of Potential Clinical Importance | |
| | | 10.6.1. | Laboratory Values | |
| | 40 = | | Vital Signs | 30 |
| | 10.7. | Appendix | 7: Model Checking and Diagnostics for Statistical | 0.4 |
| | | | Chatiatical Analysis Assumantians | |
| | 10.0 | 10.7.1. | · | |
| | 10.8. | 10.8.1. | 8: Biomarker Analyses Frequency of Leukocytes | |
| | | 10.8.1. | Frequency and phenotype of leukocyte subsets by flow | 32 |
| | | 10.0.2. | cytometry | 32 |
| | | | 10.8.2.1. B_DC_Monocyte Panel | |
| | | | 10.8.2.2. T Cell panel | |
| | | | 10.8.2.3. Treg panel | |
| | | | 10.8.2.4. Ratios of effector cells to regulatory cells | 34 |
| | | | 10.8.2.5. Suppressive activity of regulatory cells | 35 |
| | | | 10.8.2.6. General Derivations | |
| | 10.9. | Appendix | (9: Abbreviations & Trade Marks | |
| | | 10.9.1. | Abbreviations | |
| | | 10.9.2. | Trademarks | |
| | 10.10. | | 10: List of Data Displays | |
| | | 10.10.1. | Data Display Numbering | 38 |
| | | | Mock Example Shell Referencing | |
| | | | Deliverable [Priority] | |
| | | | Study Population Tables | |
| | | | Biomarker Tables | |
| | | | Safety Tables | |
| | | 10.10.7. | Biomarker Figures | 42 |


| | 203158 |
|-----------------------------------------------------------|--------|
| 10.10.8. Non-ICH Listings | 45 |
| 10.11. Appendix 11: Example Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 203158:

| Revision Chronology: | | |
|---|---|---|
| 2015N246275_00 | 11-Dec-2015 | Original |
| 2015N246275_01 | 04-Apr-2016 | Changes to the exploratory objectives, removal of LN Questionnaire, plus clarifications and corrections. |
| 2015N246275_02 | 06-Oct-2016 | Corrections to Time & Events Table and screening tests |
| 2015N246275_03 | 06-Mar-2017 | Updated text around interim analyses, change to inclusion criteria and clarifications. |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Exploratory objectives 2-5 were not evaluated due to only a limited number of cells being available to analyze, as no data has been collected these have been removed from the RAP, except for Section 2 to maintain consistency with the protocol.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the frequency and phenotype of leukocyte subsets in iLN and peripheral blood in HVs and NOT1D subjects | Absolute number and/or proportion of leukocyte subsets in iLN and peripheral blood |
| Secondary Objectives | Secondary Endpoints |
| To assess the frequency and phenotype of leukocyte subsets in iLN core biopsies and iLN fine needle aspirates in HVs and NOT1D subjects | Absolute number and/or proportion of leukocyte subsets<br>in iLN core biopsies and iLN fine needle aspirates |
| To assess the safety and tolerability of iLN biopsy as well as expectations and experience of the biopsy procedure | <ul> <li>Number of AEs and SAEs following lymph node biopsy procedure</li> <li>Descriptive data obtained by a questionnaire on the acceptability of iLN biopsy in research setting.</li> </ul> |
| Exploratory Objectives* | Exploratory Endpoints |
| To assess suppression activity of T regulatory lymphocytes from the iLN and peripheral blood in HVs and NOT1D subjects | Relative levels of T lymphocyte suppressive activity of cells from iLN and peripheral blood respectively |
| To assess the frequency of cytokine-<br>producing lymphocytes in HVs and<br>NOT1D subjects | Proportion of lymphocyte populations producing pro-<br>inflammatory and/or anti-inflammatory cytokines in iLN<br>and peripheral blood |
| To assess clonal expansion of T and B lymphocyte populations in HVs and NOT1D subjects | Comparison of TCR and BCR usage in lymphocytes in iLN and peripheral blood |
| To assess the gene expression fingerprint of auto-antigen specific lymphocytes in HVs and NOT1D subjects | Gene expression levels of sorted auto antigen stimulated T lymphocyte populations in iLN and peripheral blood |
| To assess the phenotype and transcriptomic fingerprint of stromal cells from iLN core biopsy samples in HVs and NOT1D subjects | Absolute number and/or proportion of stromal cell subsets and gene expression levels of stromal cell subsets from iLN core biopsy samples Static content of coincides and the content of content of the content |

<sup>\*</sup> The Exploratory objectives / endpoints are listed in order of priority and the conduct of any experimental assays will be dependent on the material available (i.e. number of cells obtained) from iLN biopsies and peripheral blood.

#### 2.3. Study Design



## 2.4. Statistical Hypotheses

This study is designed to explore the phenotype of immune cells in the iLN and peripheral blood (such as, but not restricted to PBMCs) of NOT1D subjects compared to HVs.

There are no formal hypotheses being tested due to the exploratory nature of the study. Primary comparisons of NOT1D subjects to HVs will be made using an estimation approach, providing point estimates and confidence intervals.

Secondary comparisons of biopsy methods will be made within NOT1D subjects and HVs using an estimation approach:

- iLN biopsies will be carried out by two related methods, fine-needle aspirate (FNA) and core biopsy sampling:
- If sufficient numbers of cells to meet the cell number requirements of the primary endpoint are obtained by both biopsy methods, the primary endpoint analysis will be carried out independently for each biopsy method, otherwise only the biopsy

- method for which sufficient numbers of cells were obtained will be used for primary analysis.
- If no meaningful differences between biopsy methods are observed, material from both biopsy methods may be pooled to meet exploratory objectives 1, 2, 3 and 4. Material from fine-needle aspirate and core biopsies will not be pooled unless supported by the comparison described above.
- If meaningful differences in the proportion of leukocyte subsets between cells derived from each biopsy method are observed, then:
  - o If sufficient number of core biopsy derived cells are available, these will be analysed for exploratory objectives 1 and 2.
  - o Fine needle aspirate derived cells will be used to meet exploratory objectives 3 and 4. If insufficient number of core biopsy derived cells are available to meet exploratory objectives 1 and 2, then fine needle aspirate derived cells may be used to meet either or both of those exploratory objectives.

A graphical representation of the comparisons are shown in Figure 1.

Figure 1 - Graphical representation of comparisons



#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

#### 3.1.1. Interim Analysis 1

A data look will be carried after the recruitment of a cohort of up to 5 HVs to determine if the quality and quantity of cells derived from either fine needle aspirate or core biopsy of the inguinal lymph node and from peripheral blood are likely to be sufficient to continue the study to meet its primary objective.

The decision rules for the study to continue are:

- Peripheral blood yields  $> 1 \times 10e^6$  cells, and
- Yield from either iLN biopsy samples  $> 1 \times 10e^6$  cells.

In addition, the data from the interim analysis will be used to explore the assumptions and feasibility of the primary statistical analysis, and may also be used for pre-programming of outputs for the final analysis.

If the decision is taken to stop the study at the interim, the full safety outputs plus listings of other collected data will be produced.

#### 3.1.2. Interim Analysis 2

An interim analysis will be carried out after the recruitment of 5 evaluable HVs and 5 evaluable NOT1D subjects. The primary purpose of this interim analysis will be to facilitate decision making and study design for a potential follow-up interventional study.

In addition, the interim analysis results would also help to enable prioritization of the exploratory assays and to facilitate the final RAP. Due to uncertainty around variability and precision, the primary analyses described in Section 7 will be performed in order to re-assess the precision of estimates for the comparisons of interest.

### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population |
| Enrolled | All participants who passed screening and entered the study | Study Population |
| Safety | Comprised of all subjects who complete any study assessment | <ul><li>Study Population</li><li>Safety</li></ul> |
| Core Biopsy | Subjects in the 'Safety' population for whom at least one lymph node core biopsy was taken | Biomarker |
| Fine needle aspirate Biopsy | Subjects in the 'Safety' population for whom at least one lymph node fine needle aspirate biopsy was taken | Biomarker |
| Biopsy | Subjects in both 'Core Biopsy' and 'fine needle aspirate biopsy' populations | Biomarker |
| Blood | Subjects in the 'Safety' population for whom one blood sample was taken for analysis of cells derived from peripheral blood. | Biomarker |
| Per Protocol | Subjects in the 'Safety' Population who were compliant with the Protocol | Biomarker |

#### NOTES:

• Please refer to Appendix 10: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP).
  - Onta will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset. This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.
- Analyses may be repeated on the Per Protocol population if deemed important.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

#### 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | ng | |
| Code Description | | Description | Order [1] |
| Α | No Treatment | No Treatment | n/a |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

| Study Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | ng |
| Code | Description | Description | Order [1] |
| 1 Healthy Volunteers | | Healthy Volunteers | 1 |
| 2 | NOT1D | NOT1D | 2 |

#### 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-biopsy assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to biopsy and used as baseline.

#### 5.3. Change from Baseline Definitions

| Definition | Reporting Details |
|------------------------|----------------------------------------------------|
| Change from Baseline | =Post-Biopsy Value – Baseline |
| % Change from Baseline | =100 x [(Post-Biopsy Value – Baseline) / Baseline] |

#### 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries and statistical analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|------------|-------------------|
| Covariates | Age, Gender, Site |

#### NOTES:

- The effect of Age/Gender will be explored if it was not possible to match all subjects by age and gender.
- The effect of site will be explored

#### **5.4.2.** Examination of Subgroups

No planned subgroups will be examined.

#### 5.5. Multicentre Studies

There are no planned adjustments made for multiple centres in this study.

#### 5.6. Multiple Comparisons and Multiplicity

There are no planned adjustments for multiple comparisons or multiplicity.

## 5.7. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Model Checking and Diagnostics for Statistical Analyses |
| 10.8 | Appendix 8: Biomarker Analyses |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the enrolled population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, will be based on GSK Core Data Standards.

The number and percent of subjects will be reported for the responses for the categorical Pre-Biopsy and Post-Biopsy lymph node questionnaire data. All questions will be listed.

Details of the planned displays are presented in Appendix 10: List of Data Displays

#### 6.1.1. Interim Analysis 1

No study population analyses will be produced for the first interim analysis.

#### 6.1.2. Interim Analysis 2

No study population analyses will be produced for the first interim analysis.

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Biomarker Analyses

#### 7.1.1. Overview of Planned Biomarker Analyses

The primary biomarker analyses will be based on the 'Safety' population, unless otherwise specified.

Between group (HV vs NOT1D) comparisons will use data from all subjects who have at least one evaluable sample from either method. Between method comparisons and analyses will only be performed in subjects who provide sufficient cells from both methods in each pairwise comparison (as shown in Figure 1).

If sufficient numbers of cells to meet the cell number requirements of the primary endpoint are obtained by both biopsy methods, the primary endpoint analysis will be carried out independently for each biopsy method, otherwise only the biopsy method for which sufficient numbers of cells were obtained will be used for primary analysis.

Details of the planned displays are presented in Appendix 10: List of Data Displays

For biomarkers that indicate a difference between methods or groups, further explanatory analyses may be carried out to explore correlations between biomarkers or the impact of covariates.

#### 7.1.1.1. Interim Analyses 1

Summary statistics and a listing for the overall cell counts will be presented.

#### 7.1.1.2. Interim Analyses 2

All primary and secondary comparisons will be presented, as detailed in Appendix 10: List of Data Displays

#### 7.1.2. Planned Biomarker Statistical Analyses

#### **Primary Statistical Analyses**

#### Endpoint(s)

Proportion of flow cytometry cell counts

#### **Model Specification**

• Endpoints analyzed for each flow cytometry cell type using generalized linear mixed models (GLMM).

The analysis will be performed on the parameters listed in

- Appendix 8: Biomarker Analyses
- Terms in GLMM model will include:

Fixed categorical: group, sample type, and the interaction of group with sample type Random effect: subject

Where group is either HV or NOT1D, and sample type is peripheral blood, core biopsy or fine needle aspirate.

#### **Model Checking & Diagnostics**

#### Refer to

Appendix 7: Model Checking and Diagnostics for Statistical Analyses

#### **Model Results Presentation**

For proportional cell counts, these models will estimate the mean (or geometric mean)
proportion for each sample type in each group, comparing means using differences or ratios as
outlined in the primary hypothesis section.

#### 7.2. Secondary statistical analyses

## 7.3. Biomarker Analyses

#### 7.3.1. Overview of Planned Biomarker Analyses

As per Primary Analysis, see Section 7.1, but for secondary comparisons detailed in Figure 1.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

#### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays

#### 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

#### 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned

#### 8.3.1. Interim Analysis 1

No formal safety analyses will be produced for the interim analysis.

#### 8.3.2. Interim Analysis 2

No formal safety analyses will be produced for the interim analysis.

#### 9. REFERENCES

GlaxoSmithKline Document Number 2015N246275\_03 (2017-MAR-06 Amendment No. 3): Exploration of the peripheral immune system in subjects with New Onset T1 Diabetes (NOT1D)

#### 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 10.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|--------|----------------------------------------|
| 01 | Eligibility criteria not met |
| 02 | Excluded medication, vaccine or device |
| 03 | Equipment procedures |
| 04 | Biological sample specimen procedures |

## 10.2. Appendix 2: Schedule of Activities

#### 10.2.1. Protocol Defined Time & Events

Screening procedures in addition to those listed below are (outpatient visit): Informed consent; Inclusion / Exclusion criteria; demography.

| Procedure | Screening (between -<br>56 to 7 days prior to<br>study session) | Study Session<br>Day 1 | | | Telephone<br>follow-up<br>Day ~2 to ~<br>Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes |
|---|---|---|---|---|---|---|---|
| | | Pre biopsy | Biopsy | End of study session visit | | | |
| Full physical exam | Х | | | | | | To be completed if a post study visit is required. Attendance to the unit post study sessions only if necessary (at discretion of investigator) |
| Medical history /<br>Past and current<br>medical conditions | X | Х | | | | | To be completed if a post study visit is required. Attendance to the unit post study sessions only if necessary (at discretion of investigator) |

| Procedure | Screening (between -<br>56 to 7 days prior to<br>study session) | Study Session<br>Day 1 | | | Telephone<br>follow-up<br>Day ~2 to ~<br>Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes |
|---|---|---|---|---|---|---|---|
| | | Pre biopsy | Biopsy | End of study session visit | | | |
| Laboratory<br>assessments | X <sup>1</sup> | <b>X</b> <sup>2</sup> | | | | | To be completed if a post study visit is required. Attendance to the unit post study sessions only if necessary (at discretion of investigator). 1. Blood testing in fasted condition at screening 2. Haematology and clinical chemistry only on Day 1 in a non fasted condition |
| Concomitant medication review | X | X | | | Х | Х | |
| Alcohol Urine Test<br>and Test for Drugs<br>of Abuse | Х | Х | | | | | |
| Urine Pregnancy<br>test (in women of<br>child bearing<br>potential) | Х | Х | | | | | |
| Procedure | Screening (between -<br>56 to 7 days prior to<br>study session) | Study Session<br>Day 1 | | | Telephone<br>follow-up<br>Day ~2 to ~<br>Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes |
|---|---|---|---|---|---|---|---|
| | , , | Pre biopsy | Biopsy | End of study session visit | | | |
| Vital signs | Х | Х | | Х | | | To be completed if a post study visit is required. Attendance to the unit post study sessions only if necessary (at discretion of investigator) |
| Proposed biopsy site review | | Х | | | | | |
| Peripheral blood collection for cell isolation | | Х | | | | | |
| Peripheral blood collection for genetics | | Х | | | | | Optional in consenting subjects |
| Inguinal lymph node<br>biopsy<br>(fine needle<br>aspirate & core<br>biopsy) | | | Х | | | | |
| Wound assessment | | | | X | X (telephone) | X<br>(telephone) | To be completed if a post study visit is required. Attendance to the unit post study sessions only if necessary (at discretion of investigator) |

| Procedure | Screening (between -<br>56 to 7 days prior to<br>study session) | Study Session<br>Day 1 | | | Telephone<br>follow-up<br>Day ~2 to ~<br>Day 4 | Telephone<br>follow-up<br>Day ~7 to<br>Day ~14 | Notes |
|---|---|---|---|---|---|---|---|
| | , | Pre biopsy | Biopsy | End of study session visit | | | |
| Pre- & post-biopsy<br>questionnaire to<br>assess subject<br>experience of lymph<br>node biopsy | | X | | | X (fill in questionnaire on the day after the procedure, communicate answers via telephone a few days after) | | |
| SAE review | <b>←</b> | | | | <del>-</del> | | |
| AE review | | <b>←</b> | | | <del>-</del> | | |

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

### 10.3.1. Reporting Process

| Software | |
|---|---|
| The currently sur | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound | : \\arprod\nocompound\mid203158 |
| | \\arwork\nocompound\mid203158 |
| Analysis Datasets | |
| Analysis datasets | Analysis datasets will be created according to Legacy GSK A&R dataset standards. |
| Generation of RTF Files | |
| RTF files will be generated for the final analysis tables only. | |

### 10.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visit | its will not be included in summary tables. |
| <ul> <li>Unscheduled visit</li> </ul> | its will not be included in figures. |
| All unscheduled v | visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data N, n, frequency, % | |

#### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### Multiple Measurements at One Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from date of biopsy :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Biopsy Date → Study Day = Ref Date Biopsy Date
  - Ref Data ≥ Biopsy Date → Study Day = Ref Date (Biopsy Date) + 1

#### 10.4.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
  - o The date of final screening will be used as the reference for the calculation.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### 10.4.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, will imputed using the following rules:
  - If value is below limit of quantification, then 0.5\*lower limit of quantification will be used
  - If the value is above upper limit of quantification, then the upper limit of quantification will be used.

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

## 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the follow-up call(s). The end of the study is defined as the last subject's last telephone call. As defined in the protocol the overall study duration for each subject will be up to 8 weeks, including the screening period.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in displays, unless otherwise specified.</li> </ul> |

## 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated using a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the listing.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 10.5.2.1. Handling of Missing Dates

Completely missing dates will remain missing, with no imputation applied.

## 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to day of biopsy and the event could possibly have occurred post-biopsy from the partial information, then the biopsy date will be assumed to be the start date.</li> <li>The AE will then be considered to start post-biopsy (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.5.2.3. Handling of Missing Data for Statistical Analysis

Missing data will remain missing with no imputation applied for the purposes of statistical analysis.

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /I | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decr | Decrease | | Increase |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

# 10.7. Appendix 7: Model Checking and Diagnostics for Statistical Analyses

### 10.7.1. Statistical Analysis Assumptions

| Endpoint(s) | • | Proportion of flow cytometry cell counts |
|-------------|---|------------------------------------------|
| Analysis | • | GLMM |

- Model assumptions will be applied, but appropriate adjustments maybe applied based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the RANDOM line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

# 10.8. Appendix 8: Biomarker Analyses

# 10.8.1. Frequency of Leukocytes

| Test Analyte | Details |
|---|---|
| Core biopsy total cell number | Total number of cells obtained from pooled core biopsies |
| Fine Needle Aspirate total cell number | Total number of cells obtained from pooled fine needle aspirates |

# 10.8.2. Frequency and phenotype of leukocyte subsets by flow cytometry

## 10.8.2.1. B\_DC\_Monocyte Panel

| Test Analyte | Details |
|---|---|
| %DC (MNC) | NONCD16hiCD3-CD19-NK-HLADR+CD14-CD16- out of mononuclear cells |
| %Myeloid DC (DC) | NONCD16hiCD3-CD19-NK- HLADR+CD14-CD16-<br>CD11C+CD123- |
| %pDC (DC) | NONCD16hiCD3-CD19-NK-HLADR+CD14-CD16-CD11C-CD123+ |
| %Plasmablast (B) | NONCD16hiCD19+CD27+CD38+ |
| %Circulating B (B) | NONCD16hiCD19+Plasmablast-CD27+lgD+ |
| %Classical B (B) | NONCD16hiCD19+Plasmablast-CD27+lgD- |
| %Double neg B (B) | NONCD16hiCD19+Plasmablast-CD27-lgD- |
| %Naïve B (B) | NONCD16hiCD19+Plasmablast-CD27-lgD+ |
| %Transitional B (B) | NONCD16hiCD19+Plasmablast-CD27-lgD+CD38+CD24+ |
| %CD56bright NK (NK) | NONCD16hiCD3-CD19- CD14- CD56hi CD16- |
| %CD56loCD16+ NK (NK) | NONCD16hiCD3-CD19- CD14- CD56lo CD16+ |
| %CD56loCD16- NK (NK) | NONCD16hiCD3-CD19- CD14- CD56lo CD16- |
| %CD56+CD16+ NK (NK) | NONCD16hiCD3-CD19- CD14- CD56+ CD16+ |
| % NK (MNC) | NONCD16hiCD3-CD19- CD14- out of mono-nuclear cells |
| %CD56bright NK (MNC) | NONCD16hiCD3-CD19- CD14- CD56h CD16-i out of mono-<br>nuclear cells |
| %CD56loCD16+ NK (MNC) | NONCD16hiCD3-CD19- CD14- CD56loCD16+ out of mono-<br>nuclear cells |
| %CD56loCD16- NK (MNC) | NONCD16hiCD3-CD19- CD14- CD56loCD16- out of mononuclear cells |
| %CD56+CD16+ NK (MNC) | NONCD16hiCD3-CD19- CD14- CD56+CD16+ out of mononuclear cells |
| %CD14+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD14+ |
| %CD14+CD16+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD14+CD16+ |
| %CD16+ monocyte (monocyte) | NONCD16hiCD3-CD19-NK-HLADR+Monocyte+CD16+ |
| %B (MNC) | NONCD16hiCD19+ out of mono-nuclear cells |

# 10.8.2.2. T Cell panel

| Test Analyte | Details |
|---|---|
| %CD8 Tn (CD8) | CD3+CD4-CD45RA+CCR7+CD95- |
| %CD8 Tcm (CD8) | CD3+CD4-CD45RA-CCR7+ |
| %CD8 Tem (CD8) | CD3+CD4-CD45RA-CCR7- |
| %CD8 Temra (CD8) | CD3+CD4-CD45RA+CCR7- |
| %CD8 Tscm (CD8) | CD3+CD4-CD45RA+CCR7+CD95+ |
| %Tconv Tn (Tconv) | CD3+CD4+Treg-CD45RA+CCR7+CD95- |
| %TconvTcm (Tconv) | CD3+CD4+Treg-CD45RA-CCR7+ |
| %Tconv Tem (Tconv) | CD3+CD4+Treg-CD45RA-CCR7- |
| %TconvTemra (Tconv) | CD3+CD4+Treg-CD45RA+CCR7- |
| %Tconv Tscm (Tconv) | CD3+CD4+Treg-CD45RA+CCR7+CD95+ |
| %Tconv Th1 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-CXCR3+CCR4-CCR10-CCR6- |
| %Tconv Th1Th17 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-CXCR3+CCR4-CCR10-CCR6+ |
| %Tconv Th1Th2 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-<br>CXCR3+CCR4+CCR10-CCR6- |
| %Tconv Th1Th17Th2 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-<br>CXCR3+CCR4+CCR10-CCR6+ |
| %TconvTh2 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-CXCR3-CCR4+CCR10-CCR6- |
| %TconvTh17 (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5-CXCR3-CCR4+CCR10-CCR6+ |
| %TconvTh22 (mTconv) | CD3+CD4+Treg-Tconv Tn- Tconv Tscm-CXCR5-CXCR3-CCR4+CCR10+CCR6+ |
| %Tconv Tfh (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5+ |
| %Tconv PD-1+ ICOS+ Tfh (mTconv) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5+PD-1+ICOS+ |
| %Treg Th1 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-CXCR3+CCR4-CCR10-CCR6- |
| %Treg Th1Th17 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-<br>CXCR3+CCR4-CCR10-CCR6+ |
| %Treg Th1Th2 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-<br>CXCR3+CCR4+CCR10-CCR6- |
| %Treg Th1Th17Th2 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-<br>CXCR3+CCR4+CCR10-CCR6+ |
| %Treg Th2 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-CXCR3-CCR4+CCR10-CCR6- |
| %Treg Th17 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-CXCR3-CCR4+CCR10-CCR6+ |

| Test Analyte | Details |
|---|---|
| %Treg Th22 (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5-CXCR3-CCR4+CCR10+CCR6+ |
| %Treg Tfh (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5+ |
| %Treg PD-1+ ICOS+ Tfh (mTreg) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5+PD-1+ICOS+ |
| %Tconv PD-1+ ICOS+ Tfh (Tconv Tfh) | CD3+CD4+Treg-Tconv Tn-Tconv Tscm-CXCR5+PD-1+ICOS+ out of Tconv Tfh |
| %Treg PD-1+ ICOS+ Tfh (Treg Tfh) | CD3+CD4+CD25+CD127loTreg Tn-Treg Tscm-CXCR5+PD-1+ICOS+ out of Treg Tfh |

# 10.8.2.3. Treg panel

| Test Analyte | Details |
|--------------------------|----------------------------------------|
| %CD15s+ Tconv (Tconv) | CD3+CD4+CD25lo-medFOXP3-CD15s+ |
| %CD69+ Tconv (Tconv) | CD3+CD4+CD25lo-medFOXP3-CD69+ |
| %Helios+ Tconv (Tconv) | CD3+CD4+CD25lo-medFOXP3-HELIOS+ |
| %Ki67+ Tconv (Tconv) | CD3+CD4+CD25lo-medFOXP3-Kl67+ |
| %CD15s+ mTconv (mTconv) | CD3+CD4+CD25lo-medFOXP3-CD45RA-CD15s+ |
| %CD69+ mTconv (mTconv) | CD3+CD4+CD25lo-medFOXP3-CD45RA-CD69+ |
| %Helios+ mTconv (mTconv) | CD3+CD4+CD25lo-medFOXP3-CD45RA-HELIOS+ |
| %Ki67+ mTconv (mTconv) | CD3+CD4+CD25lo-medFOXP3-CD45RA-Kl67+ |
| %Treg (CD4) | CD3+CD4+CD25hiFOXP3+ |
| %aTreg (Treg) | CD3+CD4+CD25hiFOXP3hiCD45RA- |
| %mTreg (Treg) | CD3+CD4+CD25hiFOXP3medCD54RA- |
| %rTreg (Treg) | CD3+CD4+CD25hiFOXP3medCD45RA+ |
| %CD15s+ Treg (Treg) | CD3+CD4+CD25hiFOXP3+CD15s+ |
| %CD69+ Treg (Treg) | CD3+CD4+CD25hiFOXP3+CD69+ |
| %Helios+ Treg (Treg) | CD3+CD4+CD25hiFOXP3+HELIOS+ |
| %Ki67+ Treg (Treg) | CD3+CD4+CD25hiFOXP3+KI67+ |
| %CD69+ CD8 (CD8) | CD3+CD8+CD69+ |
| %Ki67+ CD8 (CD8) | CD3+CD8+KI67+ |

# 10.8.2.4. Ratios of effector cells to regulatory cells

The following parameters are derived.

| Test analyte | Details |
|--------------------|---------------------------------------------------------|
| Th1 Tconv:Treg | Th1 Tconv cell to Treg cell ratio |
| | Derivation: [%Tconv Th1 (mTconv)] / [%Treg Th1 (mTreg)] |
| Th1Th17 Tconv:Treg | Th1Th17 Tconv cell to Th1Th17reg cell ratio |

| Test analyte | Details |
|---|---|
| | Derivation: [%Tconv Th1Th17 (mTconv)] / [%Treg Th1Th17 (mTreg)] |
| Th1Th2 Tconv:Treg | Th1Th2 Tconv cell to Th1Th2reg cell ratio |
| | Derivation: [%Tconv Th1Th2 (mTconv)] / [%Treg Th1Th2 (mTreg)] |
| Th1Th17Th2 Tconv:Treg | Th1Th17Th2 Tconv cell to Th1Th17Th2reg cell ratio |
| | Derivation: [%Tconv Th1Th17Th2 (mTconv)] / [%Treg Th1 h1Th17Th2 (mTreg)] |
| Th2 Tconv:Treg ratio | Th2 Tconv cell to Th2reg cell ratio |
| | Derivation: [%TconvTh2 (mTconv)] / [%Treg Th2 (mTreg)] |
| Th17 Tconv:Treg ratio | Th17 Tconv cell to T17reg cell ratio |
| | Derivation: [%TconvTh17 (mTconv)] / [%Treg Th17 (mTreg)] |
| Th22 Tconv:Treg ratio | Th22 Tconv cell to Th22reg cell ratio |
| | Derivation: [%TconvTh22 (mTconv)] / [%Treg Th22 (mTreg)] |
| Tfh Tconv:Treg ratio | Tfh Tconv cell to Tfhreg cell ratio |
| | Derivation: [%Tconv Tfh (mTconv)] / [%Treg Thfh (mTreg)] |

## 10.8.2.5. Suppressive activity of regulatory cells

| Test Analyte | Details |
|----------------------------|------------------------------------|
| Percentage suppression 0:1 | Treg: Tconventional cell ratio 0:1 |
| Percentage suppression 1:2 | Treg: Tconventional cell ratio 1:2 |
| Percentage suppression 1:4 | Treg: Tconventional cell ratio 1:4 |

## 10.8.2.6. General Derivations

For the parameters in Section 10.8.2.1, Section 10.8.2.2 and Section 10.8.2.3, the percentages will be transformed into counts by multiplying by the denominator counts / 100. The denominator counts are given in brackets in the test analyte column.

# 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| Abbreviation | Description |
|--------------|-------------------------------------------|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| BL | Baseline |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FNA | Fine needle aspirate |
| HV | Healthy volunteer |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| iLN | Inguinal lymph node |
| IMMS | International Modules Management System |
| GLMM | Generalized linear mixed model |
| GUI | Guidance |
| GSK | GlaxoSmithKline |
| NOT1D | New Onset Type 1 Diabetes Mellitus |
| PBMC | Peripheral blood mononuclear cell |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PP | Per Protocol |
| PT | Preferred Term |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SOC | System Organ Class |
| TCR / BCR | T-cell Receptor / B-cell Receptor |
| TFL | Tables, Figures & Listings |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

## 10.10. Appendix 10: List of Data Displays

## 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|--------------|
| Study Population | 1.01 to 1.nn | 1.01 to 1.nn |
| Biomarker | 2.01 to 2.nn | 2.01 to 2.nn |
| Safety | 3.01 to 3.nn | 3.01 to 3.nn |
| Section Listings | | ngs |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

## 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | SP_Fn | SP_Tn | SP_Ln |
| Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.10.3. Deliverable [Priority]

| Delivery | Description |
|----------|------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |

# 10.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Subje | ect Disposition | ) | | • | |
| 1.01 | Enrolled | ES1 | Summary of Subject Disposition | | SAC |
| 1.02 | Screened | ES6 | Summary of Screen Failures (Screened Subjects Population) | | SAC |
| 1.03 | Enrolled | NS3 | Summary of Subjects by Country and Centre | | SAC |
| Popu | lation Analyze | d | | | |
| 1.04 | Screened | SP1 | Summary of Study Populations | | SAC |
| Demo | ographic and E | Baseline Ch | aracteristics | • | |
| 1.05 | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.06 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| Curre | ent and Past M | edical Cond | ditions | | |
| 1.07 | Safety | MH4 | Summary of Past Medical Conditions | | SAC |
| 1.08 | Safety | MH4 | Summary of Current Medical Conditions | | SAC |
| Conc | omitant Medic | ations | | | |
| 1.09 | Safety | CM1 | Summary of Concomitant Medications | | SAC |
| Lymp | Lymph Node Questionnaire | | | | |
| 1.10 | Safety | SP_T1 | Summary of Pre-Biopsy Lymph<br>Node Questionnaire | | SAC |
| 1.11 | Safety | SP_T1 | Summary of Post-Biopsy Lymph<br>Node Questionnaire | | SAC |

# 10.10.5. Biomarker Tables

| Bioma | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Popula<br>tion | IDSL /<br>TST ID<br>/<br>Examp<br>le Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| Freque | ency and p | henotype | of leukocyte subsets by flow cytometry | | |
| 2.01 | Safety | PD_T1 | Summary of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 2.02 | Safety | PD_T2 | Statistical Analyses of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 2.03 | Safety | PD_T1 | Summary of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 2.04 | Safety | PD_T2 | Statistical Analyses of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 2.05 | Safety | PD_T1 | Summary of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 2.06 | Safety | PD_T2 | Statistical Analyses of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 2.07 | Safety | PD_T1 | Summary of ratios of effector cells to regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| 2.08 | Safety | PD_T2 | Statistical Analyses of ratios of effector cells to regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| Suppre | Suppressive activity of regulatory cells | | | | |
| 2.09 | Safety | PD_T1 | Summary of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |
| 2.10 | Safety | PD_T2 | Statistical Analyses of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |

# 10.10.6. Safety Tables

| Safet | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Adve | rse Events (A | Es) | | | |
| 3.01 | Safety | AE1 | Summary of Adverse Events<br>Summary by SOC and PT | | SAC |
| 3.02 | Safety | AE15 | Summary of Common (>=5% incidence) Non-Serious Adverse Events by SOC and PT (No. of Subjects and occurrences) | | SAC |
| 3.03 | Safety | AE5A | Summary of All Adverse Events by<br>Maximum Intensity by System<br>Organ Class and Preferred Term | | SAC |
| Serio | us Adverse E | vents | | | |
| 3.04 | Safety | AE16 | Summary of Serious Adverse<br>Events by SOC and PT (No. of<br>Subjects and occurrences) | | SAC |
| 3.05 | Safety | AE1 | Summary of Adverse Events<br>Leading to Withdrawal from Study<br>by SOC and PT | | SAC |
| Vital | Signs | | | | |
| 3.06 | Safety | VS1 | Summary of change from baseline in Vital Signs | | SAC |
| 3.07 | Safety | VS7 | Summary of Vital Sign Results<br>Relative to Potential Clinical<br>Importance (PCI) Criteria Post-<br>Baseline Relative to Baseline | | SAC |

# 10.10.7. Biomarker Figures

| Bioma | rker: Figu | res | | | |
|---|---|---|---|---|---|
| No. | Popula<br>tion | IDSL /<br>TST ID<br>/<br>Examp<br>le Shell | Title | Programming<br>Notes | Delivera<br>ble<br>[Priority] |
| Freque | ency and p | henotype | of leukocyte subsets by flow cytometry | | |
| 2.01 | Safety | PD_F1 | Boxplots of B_DC_Monocyte Panel by Method and Patient Group | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 2.02 | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of B_DC_Monocyte Panel | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 2.03 | Safety | PD_F1 | Boxplots of T Cell Panel by Method and Patient Group | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 2.04 | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of T Cell Panel | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 2.05 | Safety | PD_F1 | Boxplots of Treg Panel by Method and Patient Group | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 2.06 | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of Treg Panel | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 2.07 | Safety | PD_F1 | Boxplots of ratios of effector cells to regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| 2.08 | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of ratios of effector cells to regulatory cells | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| Suppr | Suppressive activity of regulatory cells | | | | |
| 2.09 | Safety | PD_F1 | Boxplots of Suppressive activity of regulatory cells by Method and Patient Group | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |
| 2.10 | Safety | PD_F2 | LS Mean Estimates and Differences with 95% CI of Suppressive activity of regulatory cells | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |

| ICH: | : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Subj | ect Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC |
| 2. | Enrolled | ES2 | Listing of Reasons for Subject<br>Withdrawal | | SAC |
| 3. | Screened | ES9 | Listing of Subjects who were rescreened | | SAC |
| Inclu | ısion / Exclusio | n Criteria | | | |
| 4. | Enrolled | IE3 | Listing of Eligibility Criteria Not Met | | SAC |
| Prot | ocol Deviations | | | | |
| 5. | Enrolled | DV2 | Listing of Important Protocol Deviations | | SAC |
| Popu | ulations Analys | ed | | | |
| 6. | Screened | SP3 | Listing of Subjects excluded from any population | | SAC |
| Dem | ographic Chara | cteristics | | | |
| 7. | Enrolled | DM2 | Listing of Demographic Characteristics | | SAC |
| 8. | Enrolled | DM9 | Listing of Race and Racial<br>Combinations | | SAC |
| Curr | ent and Past Mo | edical Cond | litions | | |
| 9. | Enrolled | MH2 | Listing of Current and Past Medical Conditions | | SAC |
| Prio | and Concomit | ant Medica | tions | | |
| 10. | Enrolled | CM3 | Listing of Concomitant Medications | | SAC |
| Adve | erse Events | | | | |
| 11. | Safety | AE8 | Listing of All Adverse Events | | SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 13. | Safety | AE8 | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | SAC |
| 14. | Safety | AE8 | Listing of Adverse Events Leading to Study Withdrawal | | SAC |
| 15. | Safety | AE14 | Listing of Reasons for considering a serious AE | | SAC |
| Labo | oratory | | | | |
| 16. | Safety | LB5 | Listing of Laboratory Results:<br>Hematology | | SAC |

| ICH: | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 17. | Safety | LB5 | Listing of Laboratory Results:<br>Clinical Chemistry | | SAC |
| 18. | Safety | UR2A | Listing of Laboratory Results:<br>Urinalysis | | SAC |
| Vital | Signs | | | | |
| 19. | Safety | VS4 | Listing of Vital Signs | | SAC |
| 20. | Safety | VS4 | Listing of All Vital Signs for<br>Subjects with any Value of<br>Potential Clinical Importance | | SAC |
| Preg | Pregnancy | | | | |
| 21. | Safety | PREG1A | Listing of subjects who became pregnant during the study | | SAC |

# 10.10.8. Non-ICH Listings

| Non | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| Biop | Biopsy Details | | | | |
| 22. | Safety | PD_L3 | Listing of Biopsy Sample Details | | SAC |
| Lym | ph Node ( | Questionnai | re | | |
| 23. | Safety | SP_L1 | Listing of Pre-Biopsy Lymph Node Questionnaire Data | | SAC |
| 24. | Safety | SP_L1 | Listing of Post-Biopsy Lymph Node Questionnaire Data | | SAC |
| Freq | uency and | d phenotype | e of leukocyte subsets by flow cytometry | | |
| 25. | Safety | PD_L1 | Listing of B_DC_Monocyte Panel by Biomarker | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 26. | Safety | PD_L2 | Listing of B_DC_Monocyte Panel by Group and Subject ID | Parameters listed in Section 10.8.2.1 | IA SAC,<br>SAC |
| 27. | Safety | PD_L1 | Listing of T Cell Panel by Biomarker | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 28. | Safety | PD_L2 | Listing of T Cell Panel by Group and Subject ID | Parameters listed in Section 10.8.2.2 | IA SAC,<br>SAC |
| 29. | Safety | PD_L1 | Listing of Treg Panel by Biomarker | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 30. | Safety | PD_L2 | Listing of Treg Panel by Group and Subject ID | Parameters listed in Section 10.8.2.3 | IA SAC,<br>SAC |
| 31. | Safety | PD_L1 | Listing of ratios of effector cells to regulatory cells by Biomarker | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| 32. | Safety | PD_L2 | Summary of ratios of effector cells to regulatory cells by Group and Subject ID | Parameters listed in Section 10.8.2.4 | IA SAC,<br>SAC |
| Sup | Suppressive activity of regulatory cells | | | | |
| 33. | Safety | PD_L1 | Listing of Suppressive activity of regulatory cells by Biomarker | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |
| 34. | Safety | PD_L2 | Listing of Suppressive activity of regulatory cells by Group and Subject ID | Parameters listed in Section 10.8.2.5 | IA SAC,<br>SAC |

# 10.11. Appendix 11: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.